CLINICAL TRIAL: NCT03064178
Title: Anticipated Versus Actual Pain Associated With Periodontal Surgery and Use of Pain Medication
Brief Title: Use of Pain Medication Following Periodontal Procedures
Status: Completed | Type: Observational
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor and Canada Research Chair, Brock University
Other Study IDs: 13-172
Record Dates: First submitted 2017-02-19; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Periodontal Diseases; Pain
Keywords: periodontal therapy; anticipated pain; experienced pain; pain medication use
MeSH Terms: conditions — Periodontal Diseases; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study had the following aims: i. to determine the relationship between anticipated pain and actual pain experienced following periodontal surgery; and ii. determine the factors that predict the amount of pain and the amount of pain medication use following periodontal surgery.

It was hypothesized that experienced pain will be significantly less than anticipated pain. It was also hypothesized that the following factors will affect pain experienced: sex, type of surgery, nervousness, anticipated pain, sedation, age, smoking status, supplement use and pain pill usage. It was hypothesized that the following factors will affect pain pill usage: sex, type of surgery, nervousness, anticipated pain, sedation, age, smoking status, supplement use, and actual pain.

DETAILED DESCRIPTION:
Patients may delay or avoid periodontal procedures because of fear of dental pain they will experience. By understanding factors that influence pain experienced, practitioners can provide potentially provide accommodations for their patients. This study investigated if anticipated pain is similar to actual pain experienced and if there are certain factors that influence the amount of pain experienced and/or pain pill usage.

Patients kept a 7 day diary in which they recorded anticipated pain (prior to periodontal surgery) and actual pain experienced for 7 days following the surgical procedure. Patients recorded their pain (anticipated and actual) using a visual analog scale (VAS). Patients also recorded daily pain medication and nutritional supplement use in the 7 day diary.

Other information recorded included factors that could influence pain experienced and pain pill use. For pain experienced, the influence of the following factors were assessed: sex, age, type of surgery, nervousness, sedation use, smoking status, anticipated pain, nutritional supplement use and pain pill use. For pain pill use, the influence of the following factors were assessed: sex, age, type of surgery, nervousness, sedation use, smoking status, anticipated pain, nutritional supplement use and pain experienced. These factors were analyzed using regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* require dental implant surgery or soft tissue graft surgery

Exclusion Criteria:

* regularly took pain medication for pre-existing health conditions
* previous implant or soft tissue graft surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from a periodontal clinic in Southern Ontario, Canada. Patients were in need of dental implant surgery or soft tissue graft surgery.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2014-05-10 (Actual); Primary Completion 2016-03-07 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Relationship between anticipated pain and actual pain experienced | 7 days
  Visual analog scale used (mm)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beaudette JR, Fritz PC, Sullivan PJ, Piccini A, Ward WE. Investigation of factors that influence pain experienced and the use of pain medication following periodontal surgery. J Clin Periodontol. 2018 May;45(5):578-585. doi: 10.1111/jcpe.12885. Epub 2018 Apr 16. PMID 29500837